CLINICAL TRIAL: NCT05991544
Title: The Effect of Training and Follow-up Given to Cancer Patients Receiving Chemotherapy According to the Neuman Systems Model
Brief Title: The Effect of Training and Follow-up Given to Cancer Patients Receiving Chemotherapy According to the Neuman Systems Model on the Development of Oral Mucositis and Perceptions of Comfort in Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Cancer
Keywords: nurse; oral Mucositis; education
MeSH Terms: conditions — Neoplasms; Stomatitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Training and Follow-up According to the Neuman Systems Model
  Interventions: Behavioral: Training and Follow-up According to the Neuman Systems Model
- Control (No Intervention): only procedure will be applied

INTERVENTIONS:
Behavioral: Training and Follow-up According to the Neuman Systems Model — Neuman Systems Model (NSM) it presents a holistic approach to patients by including physiological, spiritual, sociocultural and five major developmental variables
  Arms: Experimental

SUMMARY:
It is aimed to prevent the development of oral mucositis or to reduce the severity of developing oral mucositis with the training to be given to patients receiving chemotherapy according to the Neuman systems model.

DETAILED DESCRIPTION:
Oral mucositis is a health problem that is commonly seen in patients receiving chemotherapy and radiotherapy, which seriously affects the quality of life and comfort of patients. In the literature, the importance of nursing education in supporting patients has been emphasized, as well as controlling the side effects in patients receiving chemotherapy and systematically evaluating the side effects. The training program to be planned in this context will increase the self-efficacy of patients and their ability to cope with the disease. Studies have shown that planned health education effectively supports knowledge, increases participation in treatment processes, and reduces anxiety. Nurses use various nursing interventions such as coaching, face-to-face education programs, telephone monitoring and home care while providing training in symptom management.

Theories and models in nursing include a set of ideas about people, health-illness, and society that will guide the care of patients.

Nurses can be successful in providing holistic care only through the use of nursing models. By using these models, nursing activities are shifting from service-oriented to patient-oriented service. In addition, the basic concepts and relations between the concepts are determined, problems are defined and solutions can be developed. Neuman Systems Model (NSM), one of these models, adopts the open system approach and the concept of holistic maintenance. The model, whose reliability and scientific aspect has been tried since the day it emerged, has contributed to nursing practices and systematized the nursing care plan. NSM offers a holistic approach to patients by including psychological, physiological, spiritual, sociocultural and five major developmental variables of the individual.

Therefore, it is a suitable model to be used for nursing practices. In this study, NSM will be used in order to evaluate patients holistically and to meet their needs during the treatment process. With the planned training and follow-up to be given to cancer patients receiving chemotherapy, the patients were followed closely for 3 months, and it will provide significant benefits both for the patient and the country's economy by monitoring the development of oral mucositis or providing the management of developing oral mucositis. By preventing the development of oral mucositis, patients will have a more comfortable process and will contribute to the country's economy by preventing hospitalizations. Because oral mucositis causes pain enough to require the use of narcotic drugs and increases the need for total parenteral nutrition. This situation increases the hospital costs and harms the country's economy. The fact that oral mucositis does not develop during the chemotherapy process will allow the treatment process to be comfortable and more effective for the patient.In the light of all this information; It is aimed to prevent the development of oral mucositis or to reduce the severity of developing oral mucositis with the training to be given to patients receiving chemotherapy according to the Neuman systems model. In this direction, it is thought that the study will make a serious contribution to the literature.

ELIGIBILITY:
Inclusion Criteria:

Receiving chemotherapy treatment No mental or communication problems, Volunteering to participate in research. having internet, Having at least primary education level, Being able to use smart phone and internet. Being on treatment that causes methotrexate, Cispilatin, Cyclophoshamide, 5-fluorouracil group oral mucositis.

-

Exclusion Criteria:

lack of internet illiteracy

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Comfort Perception Scale in Oral Mucositis | 12 week
  The scale was developed in 2019 by Erden and İpek Çoban to evaluate the perception of comfort in patients with oral mucositis. The scale consists of 31 items and 2 sub-dimensions.
Oral Mucositis Grading Index: | 12 week
  Developed by the World Health Organization and
  It is a staging scale. Grade 0: No symptoms. Grade 1: Pain or erythema. Grade 2: Painful, erythema, edema or ulcer present, but the patient can take solid foods. Grade 3:
  There is pain, erythema, edema or ulcer, the patient can only take liquid foods. Grade 4: No feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan B.TURAN, Principal Investigator — Firat University; Yasemin Erdem, Principal Investigator — Erzurum Technical University; Seda Karaman, Principal Investigator — Atatatürk Üniversitesi
Locations (1):
- Atatürk university nursing faculty, Erzurum, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No